CLINICAL TRIAL: NCT05448807
Title: A Randomized Effectiveness of Phentolamine Mesylate as a Reversing Agent for Local Anesthesia in Decreasing Self- Inflicted Soft Tissue Trauma Following Local Anaesthesia Injection for Dental Procedure in Children: Randomized Clinical Trial
Brief Title: Effectiveness of Phentolamine Mesylate as a Reversing Agent for Local Anesthesia in Children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Saad Abourawash Tolba, doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 71192
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Soft Tissue Injuries
Keywords: lip biting hematoma
MeSH Terms: conditions — Soft Tissue Injuries | interventions — Phentolamine

STUDY DESIGN:
Intervention Model Description: Intervention group: they receive phentolamine mesylate (Oraverse) injection after the completion of their dental procedures with ratio 1:1 to LA in children weighed 30 kg and more while in children less than 30 kg only half of the amount of the cartridge is administrated.
  Control group: they don't receive any reversal agent or placebo after the completion of their dental procedures.
Who Masked: Participant, Outcomes Assessor
Masking Description: This research will be a double blinded study, where the patient (participant) and the statistician will be blind to the treatment groups (to avoid detection and reporting bias). Information bias, selection bias, and confounding will be avoided in this study. The operator will not be blinded to the treatment as the test group will receive a PM (Oraverse) injection while the control group will not receive a reversal agent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- participants receiving oraverse injection after local anaesthetic administration (Experimental): participants receive phentolamine mesylate (Oraverse) injection after the completion of their dental procedures with ratio 1:1 to LA in children weighed 30 kg and more while in children less than 30 kg only half of the amount of the cartridge is administrated.
  Interventions: Drug: OraVerse
- participants with no drug after local anaesthetic administration (No Intervention): participants don't receive any reversal agent or placebo after the completion of their dental procedures.

INTERVENTIONS:
Drug: OraVerse — Phentolamine mesylate is a vaso-dilator that was used for treating dermal necrosis and severe hypertension cases since 1952. It is alpha-adrenergic antagonist. Oraverse is supplied in a dose equal to the amount of LA taken in adults and children with weights more than 30 kg. While in children less than 30 kg, it is advised to use only half carpule according the manufacturer's instructions.
  Other Names: phentolamine mesylate
  Arms: participants receiving oraverse injection after local anaesthetic administration

SUMMARY:
Local anaesthesia is considered one of the most alarming and non-comfortable dental procedures for children. This goes back to the persisting effect of the local anaesthesia after finishing dental procedures. The effect of Local anaesthesia can last from 3 to 5 hours due to the presence of vasoconstrictor. The U.S Food and Drug Administration (FDA approved the use of phentolamine mesylate (Oraverse) in May 2008 to be used as a drug in reversing the numbing effect of Local anaesthesia by decreasing the time needed to restore the normal functions of the mouth

DETAILED DESCRIPTION:
Local anesthesia is the most common method for pain control during any dental procedures, but it is also one of the factors that can trigger discomfort and anxiety in children. Local anesthetics are primarily used to reversibly block action potentials that create impulse conduction along neural axons carrying sensory or motor signals. This occurs by blocking voltage-gated sodium channels. A prospective study of 320 children by College et al., (2000), reported soft tissue trauma frequency as 18%, 16%, 13% and 7% in children who are; less than 4, 4-7, 8-11 and more than 12 years old, respectively following inferior alveolar nerve block anesthesia and its numbing effect.

The search for a pharmacologic means of minimizing postoperative soft tissue anesthesia has focused on phentolamine mesylate (PM), where an injectable form has been developed. Following the administration of local anesthetic with vasoconstrictor, a subsequent phentolamine injection into the same location enhances the redistribution of the local anesthetic away from the injection site as it is an alpha-adrenergic blocking agent, explaining the more rapid return of normal intraoral and perioral sensation.

An intra-oral preparation of PM for the reversal of soft tissue anesthesia was approved by the FDA in May 2008, to be used for patients > 6 years of age and weighing > 15 kg. Later, in March 2016, the FDA approved its use in pediatric patients 3 years and older. Dosage form of OraVerse (phentolamine mesylate) is 0.4 mg/1.7 ml solution per cartridge. Its maximum dose is 2 cartridges in adults. The first published placebo-controlled phase two study reported that, in 10- to 58-year-old dental patients, an injection of phentolamine, at a one-to-one ratio at the site of the previous injection of local anesthesia, accelerated median recovery time to normal sensation of the upper and lower lips by 85 minutes.

ELIGIBILITY:
Inclusion Criteria:

Children aged 5-7 years.

* Patients in need of dental procedures requiring local anaesthesia.
* Healthy Children without any systemic or mental disorders.
* Normal lip sensation before administration of LA.
* Normal paediatric functional assessment battery (pFAB) for smiling, speaking and drinking and absence of drooling.

Exclusion Criteria:

* Children seeking dental treatment that does not necessitate local anaesthesia.
* Children who didn't achieve profound numbness requiring additional anaesthesia.
* Children who lack the ability to distinct the anaesthetised numb side from the non-anaesthetised one.
* Children who are not willing to participate in the study.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-07-05 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time to return to normal function | 2 hours
  it is the time needed for the soft intraoral tisues e.g lips, tongue to return to their normal functions after local anaesthesia

SECONDARY OUTCOMES:
Incidence of self-inflicted soft tissue trauma | 2 hours
  we observe clinical signs of redness, swelling, hematoma or ulcers due to lip biting at dismal of each participant
Cost effectiveness of oraverse | Through the completion of the study, with average 1 year
  we measure the cost effectiveness of the intervention drug through Incremental cost-effectiveness ratio (ICER) ICER=(C1-C0)/ (E1-E0) C1= cost of intervention drug C0= cost of control E1= effect of intervention drug E0= effect of control
post-operative pain by 170 mm Heft-parker visual analogue scale (VAS) | the following 24 hours
  it is 170mm scale from 0 to 170 mm and it represents
  * no pain: corresponds to 0 mm.
  * mild pain: greater than 0 mm and less than or equal to 54 mm and included the description of faint and weak pain.
  * moderate pain: greater than 54 mm and less than 114 mm.
  * severe pain: equal to or greater than 114 mm to 170 mm and includes the description of strong and intense pain

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud hamdy, professor, Study Chair — main supervisor
Locations (1):
- Cairo University, Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No